CLINICAL TRIAL: NCT04115540
Title: Transcutaneous Electrical Nerve Stimulation of Penile Nerves for Treatment of Delayed Ejaculation
Brief Title: Penile Nerve Stimulation for Treatment of Delayed Ejaculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Eisenberg, Associate Professor of Urology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52213
Record Dates: First submitted 2019-09-30; First posted 2019-10-04 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Delayed Ejaculation
MeSH Terms: conditions — Ejaculatory Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TENS penile nerve stimulation group (Experimental): The electrode pads of the transcutaneous electrical nerve stimulation (TENS 7000) will be placed at the base of the penis (and perineum). Participants will be able to use the device prior to sexual activity (immediately before sexual encounter for 10 minutes or daily for up to 14 days prior) to "prime" their system or during sexual activity. Each participant will use the device these three separate ways for 6 weeks each (total of 18 weeks of use).
  Interventions: Device: TENS penile nerve stimulation

INTERVENTIONS:
Device: TENS penile nerve stimulation — The electrode pads of the transcutaneous electrical nerve stimulation (TENS 7000) will be placed at the base of the penis (and perineum) to stimulate the penile nerves.

SUMMARY:
The aim of this clinical trial is to test the safety and feasibility of using transcutaneous electrical nerve stimulation (TENS) of the penile nerves to reduce intra-vaginal ejaculatory latency time in men with delayed ejaculation (DE). We hypothesize that this type of stimulation, either before or during sexual activity, will reduce latency time. The primary objective of this study is to determine if TENS of the penile nerve helps men with DE subjectively reduce their ejaculatory latency time. The secondary objective is to determine whether their International Index of Erectile Function (IIEF) score improves with treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Sexually active
* Diagnosed with delayed ejaculation

Exclusion Criteria:

* Less than 18 years old
* Any condition effecting the participant that would make them unable to operate the interventional device

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eisenberg, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Healthcare, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and study protocol set will be available upon request from the authors.
Supporting Information: Study Protocol
Time Frame: Data will be made available after publication of the study results for at least 3 years.

RESULTS

PARTICIPANT FLOW:
Groups:
- TENS Penile Nerve Stimulation Group: Electrode pads of the transcutaneous electrical nerve stimulation (TENS 7000) placed on the penis to stimulate the penile nerves.
Period: Overall Study
Arm/Group | TENS Penile Nerve Stimulation Group
Started | 20
Completed | 6
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | TENS Penile Nerve Stimulation Group
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12
  Asian | 1
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: International Index of Erectile Function (IIEF) Scale Score
Description: Participants were surveyed before testing the device and then at the conclusion of the trial using the International Index of Erectile Function (IIEF) which is a validated multidimensional scale for erectile function and ejaculatory function in men. The questionnaire consists of 3 questions with a scale for each from 0-5 (highest overall score 15, lowest score 0). The higher the score, the better the outcome and vice versa.
Time Frame: Baseline and 12 weeks
Population: Participants with data at baseline and week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENS Penile Nerve Stimulation Group
Number analyzed (Participants) | 6
score on a scale
  Baseline | 7.5 (4.6)
  Week 12 | 9.7 (2.2)

2. Secondary Outcome: Count of Participants With Treatment-related Adverse Events as Assessed by Survey
Description: Participants were asked about treatment related adverse events via Qualtrics survey at the conclusion of the study.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TENS Penile Nerve Stimulation Group
Number analyzed (Participants) | 14
Participants | 0

3. Post Hoc Outcome: Overall Satisfaction Scale Score
Description: The questionnaire consists of 2 questions with a scale for each from 0-5 (highest overall score 10, lowest score 0). The higher the score, the better the satisfaction and vice versa.
Time Frame: Baseline and 12 weeks
Population: Participants with data at baseline and week 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENS Penile Nerve Stimulation Group
Number analyzed (Participants) | 6
score on a scale
  Baseline | 6.0 (3.0)
  Week 12 | 7.8 (1.0)

4. Post Hoc Outcome: Number of Participants With Symptom Improvement
Description: Participants were asked yes/no questions regarding improvement in sexual activity
Time Frame: 12 weeks
Population: Participants who completed the protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TENS Penile Nerve Stimulation Group
Number analyzed (Participants) | 6
Participants
  Improved sexual activity | 4
  Able to ejaculate faster | 3
  Able to ejaculate more often | 2

5. Post Hoc Outcome: Number of Participants Utilizing TENS Prior to Intercourse, During Intercourse, and Daily
Time Frame: 12 weeks
Population: Participants who reported data for the respective questions
Measure: Count of Participants; unit: Participants
Arm/Group | TENS Penile Nerve Stimulation Group
Number analyzed (Participants) | 14
Participants
  During sexual activity | 5
  Before sexual activity: number analyzed (Participants) | 9
  Before sexual activity | 3
  Daily use: number analyzed (Participants) | 8
  Daily use | 3

6. Post Hoc Outcome: Number of Participants With Device-related Pain
Description: Device related pain would not necessarily be considered to be an adverse event
Time Frame: 12 weeks
Population: Participants who completed the protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TENS Penile Nerve Stimulation Group
Number analyzed (Participants) | 6
Participants | 2

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | TENS Penile Nerve Stimulation Group
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT04115540/Prot_001.pdf